CLINICAL TRIAL: NCT00349063
Title: The Impact of Short Term Wearing Time on In Vivo and Ex Vivo Wettability
Brief Title: Contact Lens Wettability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P/217/05/L
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors | interventions — Contact Lenses, Hydrophilic

INTERVENTIONS:
Device: soft contact lens
Drug: Soft contact lens multipurpose disinfection regimen

SUMMARY:
The purpose of this study is to compare the wettability of contact lenses disinfected with three marketed contact lens care solutions.

ELIGIBILITY:
Inclusion Criteria:

1. Has had an oculo-visual examination in the last two years.
2. Is at least 18 years old and has full legal capacity to volunteer or is at least 16 years old, has a parent or guardian's permission to participate in the study and has read the Information and Consent Letter for adolescents.

4. Has read and understood the Information Consent Letter (Appendix II). 5. Is willing and able to follow participant instructions for product usage and meet the protocol-specified schedule of follow-up visits.

6. Has a refractive error that is correctable with the prescription of the available study lenses.

7. Has a refractive error that is correctable to at least 20/25 distance visual acuity with contact lenses in each eye.

8. Has acceptable fit with the study lenses. 9. Has clear corneas, and ocular clinical findings are considered "normal".

Exclusion Criteria:

1. Has any systemic disease that may affect ocular health.
2. Is using any systemic or topical medications that may affect ocular health.
3. Has any ocular pathology or severe insufficiency of lacrimal secretion (dry eyes) that may affect the wearing of contact lenses.
4. Has any clinically significant lid or conjunctival abnormalities, meibomian gland dysfunction, neovascularization, corneal scars or corneal opacities.
5. Has limbal injection, bulbar injection or corneal staining that, in the investigator's opinion, is clinically significant.
6. Has pinguecula and/or pterygium that, in the investigator's judgement, makes contact lens wear inadvisable.
7. Has refractive astigmatism of more than 0.75 D.
8. Has corneal distortion resulting from rigid lens wear.
9. Is aphakic.
10. Has undergone corneal refractive surgery.
11. Is participating in any other type of clinical or research study.
12. Is pregnant or lactating.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 55
Dates: Start 2005-07

PRIMARY OUTCOMES:
To investigate the impact of wearing time and contact lens care solutions on in
vivo and ex vivo wettability of currently marketed contact lenses

SECONDARY OUTCOMES:
To determine if there is a correlation between in vivo wettability, ex vivo
wettability and in-eye comfort. To determine if comfort and wettability vary
between symptomatic and asymptomatic lens wearers.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Woods, PhD, Principal Investigator — University of Waterloo; Desmond Fonn, MOptom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada